CLINICAL TRIAL: NCT03564392
Title: The Investigation of a Remotely Delivered Behavioral Intervention for Postoperative Weight Regain
Brief Title: Post-Bariatric Weight Regain Behavioral Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Lauren Bradley, Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16062305
Record Dates: First submitted 2018-04-26; First posted 2018-06-20 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Ten weekly modules will be delivered through an e-learning platform (i.e., Coursesites). Each module includes a video presentation of material synchronized with a slideshow illustrating session material with interactive features, and directed assignments to be completed throughout the week. At the end of every two weeks, a brief (i.e., 20 min) telephone call with a member of the study team will be scheduled to discuss and clarify the content of the session, discuss how the participant utilized skills demonstrated in the session, problem-solve difficulties in utilizing the skills, and review homework. Participants will be required to weigh themselves weekly (data will be transferred wirelessly to the laboratory) and feedback regarding weight losses will be provided during the phone call. The interventionist will provide individualized feedback on food records via email.
  Interventions: Behavioral: Acceptance Based Behavioral Intervention
- Wait List Control (No Intervention): The Wait-List Control (WLC) condition does not receive any intervention during the study period. They receive the intervention after completing the study.

INTERVENTIONS:
Behavioral: Acceptance Based Behavioral Intervention — This intervention focuses on acceptance-based strategies with an emphasis on willingness to experience less pleasurable internal experiences (e.g., pleasure from eating calorically-dense foods) and aversive internal experiences (e.g., hunger, food cravings). Strategies to increase this willingness will be taught, including defusion (i.e., getting psychological distance from internal experiences to allow oneself to act independently of them). Mindful decision-making, as it relates to eating and exercise, will also be emphasized. Clarification and commitment to core values is another key component, as living life in accordance with one's values (e.g., health) makes willingness to make difficult choices worthwhile. Standard behavioral techniques for weight loss (i.e., self-monitoring, stimulus control, psychoeducation) will also be included.
  Arms: Treatment

SUMMARY:
This project aims to evaluate a newly developed Internet-delivered (via e-learning modules) acceptance-based behavioral intervention (ABTi) for individuals who are experiencing weight regain after bariatric surgery. Specifically, the investigators aim to assess ABTi's efficacy on stopping and/or reversing weight by comparing it to a wait-list control (WLC) condition. The investigators also aim to evaluate its effect on targeted weight control behaviors and acceptance-based skills. Finally, the investigators will examine the relationship between weight outcomes and changes in process variables through exploratory analyses. Treatment outcomes (i.e., weight, maladaptive behaviors, physical activity, acceptance-based skills) will be measured at assessments pre-, mid-, and post-treatment, as well as at 3 months after treatment has ended.

Primary Aims.

1. To test the hypothesis that participants randomly assigned to ABTi will display greater weight loss from pre- to post-treatment than those assigned to WLC.
2. To test the hypothesis those receiving ABTi, compared to WLC, will display decreased maladaptive eating behaviors (i.e., loss of control episodes, grazing, emotional eating, disinhibition), increased physical activity, and greater improvements in acceptance-based skills (i.e., mindfulness, defusion, food-related acceptance).

Exploratory Aim.

(1) To assess if changes in acceptance-based skills, maladaptive eating behaviors, and physical activity are associated with pre- to post-treatment weight outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone any type of weight loss surgery at least 1.5 years ago
* Demonstrate ≥ 10% weight regain of maximum weight loss or 5% of their minimum weight post-surgery, with weight regain lasting for at least 3 months prior to enrollment.
* Ability to give consent and speak, write, and understand English.

Exclusion Criteria:

* Currently enrolled in structured weight loss program
* Currently pregnant/plan to become pregnant within 6 months of enrollment
* Have a serious medical condition that has the potential of affecting weight or that would prevent engagement in dietary changes and/or an exercise regimen
* Exhibit psychiatric symptoms that would interfere with the ability to benefit from the intervention, or report acute suicidality
* Non-ambulatory (i.e., unable to walk at least one city block without a cane or walker at the time of screening
* Use of medications known to affect body weight, such as chronic systemic steroids or psychiatric medications including lithium, tricyclic antidepressants, and antipsychotic agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Weight loss | 10 weeks

SECONDARY OUTCOMES:
Loss of Control Eating Scale (LOCES) | 10 weeks
  LOCES measures loss of control eating.
Repetitive Eating Assessment-Questionnaire (Rep(eat)) | 10 weeks
  Rep(eat) measures grazing behaviors.
Emotional Eating Scale (EES) | 10 weeks
  EES will be used to measure emotional eating
The Eating Inventory | 10 weeks
  The Eating Inventory will be used to measure disinhibition.
Paffenbarger Physical Activity Recall | 10 weeks
  Paffenbarger will be used to measure physical activity engagement
Philadelphia Mindfulness Scale (PHLMS) | 10 weeks
  PHLMS will be used to measure mindfulness
Drexel Defusion Scale (DDS) | 10 weeks
  DDS will be used to measure delusion (a psychological construct of cognitive distancing)
Food-Related Acceptance and Action Questionnaire (FAAQ) | 10 weeks
  FAAQ will be used to measure food-related acceptance

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided